CLINICAL TRIAL: NCT06293040
Title: The Impact of Vaporized Cannabis Administration and Co-Administration of Alcohol on Impairment
Brief Title: Vaporized Cannabis Administration and Co-Administration of Alcohol on Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00434441; R01DA052295 (NIH)
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cannabis Intoxication; Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — nabiximols; Dronabinol; Ethanol

STUDY DESIGN:
Intervention Model Description: All participants will complete all dose conditions (study arms) in a randomized order
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double-blind (Participant, Outcomes Assessor), placebo controlled, and double-dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo cannabis + placebo alcohol (Placebo Comparator): Participants administer vaporized cannabis containing 0mg THC in combination with a placebo alcohol drink.
  Interventions: Drug: Placebo Cannabis; Drug: Placebo Alcohol
- Low dose cannabis with placebo alcohol (Experimental): Participants administer vaporized cannabis containing 5mg THC in combination with a placebo alcohol drink.
  Interventions: Drug: Cannabis; Drug: Placebo Alcohol
- High dose cannabis with placebo alcohol (Experimental): Participants administer vaporized cannabis containing 25mg THC in combination with a placebo alcohol drink.
  Interventions: Drug: Cannabis; Drug: Placebo Alcohol
- Low dose cannabis with low dose alcohol (Experimental): Participants administer vaporized cannabis containing 5mg THC in combination with an alcohol drink (0.05 percent BAC).
  Interventions: Drug: Cannabis; Drug: Alcohol
- High dose cannabis with low dose alcohol (Experimental): Participants administer vaporized cannabis containing 25mg THC in combination with an alcohol drink (0.05 percent BAC).
  Interventions: Drug: Cannabis; Drug: Alcohol
- Placebo cannabis + low dose alcohol (Experimental): Participants administer vaporized cannabis containing 0mg THC in combination with an alcohol drink (0.05 percent BAC).
  Interventions: Drug: Alcohol; Drug: Placebo Cannabis
- Placebo cannabis + high dose alcohol (Experimental): Participants administer vaporized cannabis containing 0mg THC in combination with an alcohol drink (0.08 percent BAC).
  Interventions: Drug: Alcohol; Drug: Placebo Cannabis

INTERVENTIONS:
Drug: Cannabis — Cannabis will be vaporized using the Mighty Medic
  Other Names: THC
  Arms: High dose cannabis with low dose alcohol; High dose cannabis with placebo alcohol; Low dose cannabis with low dose alcohol; Low dose cannabis with placebo alcohol
Drug: Alcohol — Alcohol will be orally ingested via a flavored drink
  Other Names: Ethanol
  Arms: High dose cannabis with low dose alcohol; Low dose cannabis with low dose alcohol; Placebo cannabis + high dose alcohol; Placebo cannabis + low dose alcohol
Drug: Placebo Cannabis — Placebo cannabis (i.e., water vapor) will be vaporized using the Mighty Medic.
  Other Names: Placebo
  Arms: Placebo cannabis + high dose alcohol; Placebo cannabis + low dose alcohol; Placebo cannabis + placebo alcohol
Drug: Placebo Alcohol — A non-alcoholic, placebo, flavored drink will be orally ingested.
  Other Names: Placebo
  Arms: High dose cannabis with placebo alcohol; Low dose cannabis with placebo alcohol; Placebo cannabis + placebo alcohol

SUMMARY:
This human laboratory study will use cognitive, behavioral, and subjective measures to characterize impairment associated with co-use of alcohol and vaporized cannabis. Participants (n=32) will complete 7 double-blind, double-dummy outpatient sessions in randomized order. In each session, participants will self-administer placebo (0 mg THC) or active vaporized cannabis (5 or 25 mg THC, via a handheld vaporizer called the Mighty Medic) and a placebo drink (BAC 0.0%) or alcohol drink calculated to produce a breath alcohol concentration (BAC) of 0.05%. Participants will also complete a positive control session in which the participant administers placebo cannabis and alcohol at a target BAC of 0.08% (the legal threshold for driving impairment in most U.S. states).

DETAILED DESCRIPTION:
This study will be conducted at the Johns Hopkins Behavioral Pharmacology Research Unit (BPRU). Participants will complete a screening visit, and, if eligible, will then complete 7 experimental drug administration sessions in randomized order where the participant will vaporize cannabis-containing capsules (or "pods") (containing 0, 5, or 25mg THC) with a drink that contains no alcohol or alcohol (alcohol-containing drinks will be calculated to produce a breath alcohol concentration, BAC, of 0.05%). There is also a positive control session where participants will vaporize placebo cannabis with an alcohol drink calculated to produce a BAC of 0.08%. Each session will last approximately 8 hours and will be separated by at least 48 hours to allow for sufficient drug washout. Participants may complete up to 2 sessions per week. Drugs will be administered in a double-blind and double-dummy fashion (i.e., participants will always receive both active or placebo cannabis and active or placebo alcohol). During each session, a battery of assessments including blood collection, subjective questionnaire administration, cognitive performance testing, and simulated driving will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be at least 21 years of age
3. Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
4. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at each study visit
5. Have not donated blood in the prior 30 days
6. Report at least 1 day of binge drinking in the past 3 months (greater than 4 or 5 drinks on a single occasion for women and men, respectively)
7. Report at least 1 use of cannabis in the past 3 years
8. Provide negative urine test for illicit drug use (excluding THC) and negative breath alcohol test (0% BAC) at screening and before study sessions
9. Report at least 1 lifetime instance of simultaneous alcohol and cannabis use
10. Current concomitant prescription medication use that may interact with the investigational study drug, including inhibitors and inducers of CYP2CP and CYP3A4 as well as highly-protein bound drugs and drugs with a narrow therapeutic index such as warfarin, cyclosporine, and amphotericin B

Exclusion Criteria:

1. Psychoactive drug use (aside from cannabis, nicotine, alcohol, or caffeine) in the past month
2. History of or current evidence of significant medical condition that would put the participant at risk
3. Evidence of current psychiatric condition (MINI for DSM-V)
4. Meet criteria for severe alcohol use disorder (MINI for DSM-V)
5. CIWA-Ar score > 9
6. Use of cannabis, on average, more than 3 days/week over past 3 months
7. Enrollment in another clinical trial or receiving of any drug as part of research within past 30 days
8. Shipley vocabulary score <18 (corresponds to 5th grade reading level)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
DRUID application global impairment score | Up to 6 hours
  Acute cognitive and behavioral impairment will be assessed with global impairment score (range 0-100) on the DRUID app (higher scores indicate greater impairment).
Correct Trials on Paced Auditory Serial Addition Task (PASAT) | Up to 6 hours
  Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. Will report the total correct trials out of 90 recorded (lower scores indicate worse performance). Score ranges from 0-90, with 0 representing no correct trials and 90 representing 100% correct trials.
Correct Trials on the Digit Symbol Substitution Task (DSST) | Up to 6 hours
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Will report the total correct trials in 90 seconds (lower scores indicate worse performance). There is no maximum score, with a score of 0 representing either no trials completed or no correct trials. The score reflects the number of correct trials.
Cumulative score on Field Sobriety Tests | Up to 6 hours
  Impairment will be assessed using a battery of standard field sobriety tests including: the Horizontal Gaze Nystagmus Test (HGN), the Walk and Turn, the One Leg Stand, and the Modified Romberg Balance. The cumulative amount of clues observed across these tasks (out of a possible 22 clues) will be reported.
Drug Effect Questionnaire (DEQ) - Feel Drug Effect | Up to 6 hours
  The DEQ will be used to obtain subjective ratings of "feel drug effects". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire (DEQ) - Feel High | Up to 6 hours
  The DEQ will be used to obtain subjective ratings of "feel high". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire (DEQ) - Confidence to Drive | Up to 6 hours
  The DEQ will be used to obtain subjective ratings of "confidence to drive". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire (DEQ) - Willingness to Drive | Up to 6 hours
  The DEQ will be used to obtain subjective ratings of "willingness to drive". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Biphasic alcohol effects scale (BAES) - Sedative Score | Up to 6 hours
  The BAES is used to assess sedative and stimulant subjective effects of alcohol. There are 7 sedative-related questionnaire items, each presented on a scale of 0 (not at all) to 10 (extremely), which are integrated to produce an overall sedative score (0-70).
Biphasic alcohol effects scale (BAES) - Stimulant Score | Up to 6 hours
  The BAES is used to assess sedative and stimulant subjective effects of alcohol. There are 7 stimulant-related questionnaire items, each presented on a scale of 0 (not at all) to 10 (extremely), which are integrated to produce an overall stimulant score (0-70).
Subjective high assessment scale (SHAS) | Up to 6 hours
  For the SHAS, participants are presented with 13 questionnaire items, displayed on a visual analog scale anchored from 0 (normal) to 10 (extremely), which assess subjective effects of alcohol. These items are integrated to produce an overall SHAS score (0-130)
Driving performance as assessed by standard deviation of lateral position (SDLP) | Up to 6 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. SDLP (measured in cm) will be determined during each drive. This measure is a composite index of lateral control and incorporates lane weaving, swerving, and over-correcting. SDLP is the gold standard of quantifying the magnitude of driving impairment from drugs and alcohol and has excellent predictive validity to actual driving. Scores range from 0 to no upper limit. Higher scores represent higher magnitude of driving impairment.
Driving performance as assessed by composite drive score | Up to 6 hours
  Driving impairment will be assessed via a composite drive score (higher scores indicate greater impairment). The composite drive score is derived by integrating various driving outcomes. There is no upper or lower limit to possible scores.

SECONDARY OUTCOMES:
Driving performance as assessed by standard deviation of speed (SDSP) | Up to 6 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. SDSP will be determined during each drive; this measure quantifies the variability in speed (in MPH) observed.
Driving performance (mean speed) | Up to 6 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. Mean speed (in MPH) over the course of each drive will be determined.
Driving performance (number of speed exceedances) | Up to 6 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. The cumulative number of times participants exceed the allowable speed limit during each drive.
Driving performance (number of accidents) | Up to 6 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. The cumulative number of accidents (including car collisions, pedestrians hit, etc.) during each drive.
Driving performance (total rule violations) | Up to 6 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. The cumulative number of rule violations (including number of missed stop signs, illegal turns, speed exceedances, etc.) during each drive.
Driving performance (distance to lead vehicles) | Up to 6 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. The mean distance (in meters) maintained to lead vehicles during car-following segments of each drive.
Attempted Trials on the Digit Symbol Substitution Task (DSST) | Up to 6 hours
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. The number of attempted trials will be recorded
Percentage Correct on attempted trials on the Digit Symbol Substitution Task (DSST) | Up to 6 hours
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Percentage of correct trials out of those attempted will be recorded
Reaction time on Paced Auditory Serial Addition Task | Up to 6 hours
  Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. The mean reaction time (in milliseconds) to select correct responses will be recorded.
Field Sobriety Test - Score on Horizontal Gaze Nystagmus Test | Up to 6 hours
  Impairment will be assessed using performance on the Horizontal Gaze Nystagmus Test (HGN). Total score will be recorded (out of possible 6 clues, score ranges from 0-6) with higher scores indicating higher impairment.
Field Sobriety Test - Score on Walk and Turn test | Up to 6 hours
  Impairment will be assessed using performance on the the Walk and Turn. Total score will be recorded (out of a possible 8 clues, score ranges from 0-8) with higher scores indicating higher impairment.
Field Sobriety Test - Score on One Leg Stand | Up to 6 hours
  Impairment will be assessed using performance on the One Leg Stand test. Total score will be recorded (out of a possible 4 clues, score ranges from 0-4) with higher scores indicating higher impairment.
Field Sobriety Test - Score on Modified Romberg Balance | Up to 6 hours
  Impairment will be assessed using performance on the Modified Romberg Balance test. Total score will be recorded (out of a possible 4 clues, score ranges from 0-4)) with higher scores indicating higher impairment.
Drug Effect Questionnaire - Like Drug Effect | Up to 6 hours
  The DEQ will be used to obtain subjective ratings of "like drug effect". Scores range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Want more | Up to 6 hours
  The DEQ will be used to obtain subjective ratings of "want more". Scores range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Dislike Drug Effect | Up to 6 hours
  The DEQ will be used to obtain subjective ratings of "dislike drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Pharmacokinetics - CMax for THC and THC metabolites | Up to 6 hours
  Whole blood concentrations of THC, 11-OH- THC, and THCCOOH will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentration (Cmax) is determined as the highest concentration reached for each individual. Characterizing these cannabinoids will allow for adequate control for individual differences in drug absorption and metabolism in statistical analyses and assist with interpretation of subjective and behavioral outcomes.
Pharmacokinetics - AUC for THC and THC metabolites | Up to 6 hours
  Whole blood concentrations of THC, 11-OH- THC, and THCCOOH will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline. Characterizing these cannabinoids will allow for adequate control for individual differences in drug absorption and metabolism in statistical analyses and assist with interpretation of subjective and behavioral outcomes.
Pharmacokinetics - Breath Alcohol Concentration (BAC) | Up to 6 hours
  BAC will be measured using the Alco-Sensor IV. Measuring BAC is needed to confirm that participants reached the targeted BAC for a given session and to confirm adherence to pre-session alcohol abstinence requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Tory Spindle, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No